CLINICAL TRIAL: NCT03619772
Title: Altering Activation Patterns With EMG Training in the Distal Upper Extremity After Stroke
Brief Title: EMG Training for Altering Activation Patterns After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: North Carolina State University (Other); Marquette University (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Elliot Roth, Medical Director, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00206747
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Weakness, Muscle; Coordination Lack
Keywords: hand; stroke; therapy; rehabilitation
MeSH Terms: conditions — Stroke; Muscle Weakness; Ataxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral (Experimental): Participants will control game using EMG from both upper limbs.
  Interventions: Other: Bilateral
- Unilateral (Active Comparator): Participants will control game using the more impaired upper limb.
  Interventions: Other: Unilateral

INTERVENTIONS:
Other: Bilateral — Participants will control game using EMG from both upper limbs.
  Arms: Bilateral
Other: Unilateral — Participants will control game using EMG from the more impaired upper limb.
  Arms: Unilateral

SUMMARY:
Evaluation of a new EMG controlled game to improve hand function in chronic stroke survivors.

DETAILED DESCRIPTION:
Increased impairment of the hand is commonly reported as an outcome occurring after a stroke. This impairment is due mainly to the decreased ability to modulate appropriate muscle activation patterns. Issues with appropriately modifying activation patterns can profoundly affect tasks of daily living. This study is evaluating a novel software focusing on retraining hand muscle activation patterns through an Electromyographic (EMG) controlled game. Stroke survivors with chronic, severe hemiparesis of the hand will participate in a longitudinal study consisting of 3 weeks of training. We hypothesize that stroke survivors will experience a decrease in time to complete a test of EMG control, as well as improvement in hand motor control.

ELIGIBILITY:
Inclusion Criteria:

* Single, unilateral stroke at least 6 months prior to enrollment
* Moderate hand impairment defined by Stage 4 or Stage 5 on the Chedoke McMaster Stroke Assessment Scale

Exclusion Criteria:

* Visual neglect or deficits (with inability to compensate)
* Upper extremity orthopedic conditions that interfere with movement
* Cerebellar stroke

Children, prisoners, or adult unable to provide consent will not be recruited. As the procedures pose no increased risk for pregnant women, we will not specifically exclude them.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean completion time for timed test | Baseline and 3 weeks (immediately post intervention)
  Time to complete movement to 16 randomized targets

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Roth, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seo NJ, Barry A, Ghassemi M, Triandafilou KM, Stoykov ME, Vidakovic L, Roth E, Kamper DG. Use of an EMG-Controlled Game as a Therapeutic Tool to Retrain Hand Muscle Activation Patterns Following Stroke: A Pilot Study. J Neurol Phys Ther. 2022 Jul 1;46(3):198-205. doi: 10.1097/NPT.0000000000000398. Epub 2022 Mar 22. PMID 35320135